CLINICAL TRIAL: NCT06384144
Title: Machine Learning Miscarriage Management Clinical Decision Support Tool Study
Acronym: MLMM
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 23QC8155
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Miscarriage in First Trimester

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Expectant Management of Miscarriage: Cohort that chose to pursue expectant management of miscarriage, final outcome success or failure by day 14 from management choice
  Interventions: Other: Expectant Management of First Trimester Miscarriage
- Medical Management of Miscarriage: Cohort that chose to pursue medical management of miscarriage, final outcome success or failure by day 14 from management choice
  Interventions: Other: Medical Management of First Trimester Miscarriage

INTERVENTIONS:
Other: Expectant Management of First Trimester Miscarriage — Expectant Management: Conservative management if miscarriage with follow-up booked in 2 weeks to determine whether complete miscarriage has occurred.
  Groups: Expectant Management of Miscarriage
Other: Medical Management of First Trimester Miscarriage — Medical Management: Misoprostol taken to manage first trimester miscarriage, with follow-up booked in 2 weeks to determine whether complete miscarriage has occurred.
  Groups: Medical Management of Miscarriage

SUMMARY:
Machine learning used to develop an algorithm to determine chance of success with expectant or medical management for an individual patient. Taking into account the following objective measures:

* Demographics: Maternal Age, Parity
* History: Previous CS, Previous SMM/MVA, Previous Myomectomy
* Gestation by LMP
* Presenting symptoms: Bleeding score, Pain score
* USS Measurements: CRL, GS, RPOC 3 dimensions, Vascularity
* Discrepancy between gestation by CRL and LMP

Audit to collate 1000 cases and identify features contributing to an algorithm that can predict outcome of miscarriage management for individualized case management.

DETAILED DESCRIPTION:
* Artificial intelligence discovery science: Algorithm Development based on a retrospective Audit of approximately 1000 cases of miscarriage
* To determine the reliability of the tool with test data sets
* To increase the sensitivity and specificity of the decision aid by widening the data collection to multiple sites and testing the algorithm with prospective data

The study will be conducted at Queen Charlotte's and Chelsea Hospital at Imperial College Healthcare NHS Trusts (Primary Centre of the study).

This is a multi-centre retrospective, cohort observational study.

The study will be conducted over a minimum of three years to enable sufficient time to go through the retrospective data and collate test data sets.

Retrospective annonymised cases of missed miscarriage and incomplete miscarriage managed at Imperial College Healthcare NHS Trust will be analyse:

For each case the following clinical features will be collated and outcomes:

* Demographics: Maternal Age, Parity
* History: Previous CS, Previous SMM/MVA, Previous Myomectomy
* Gestation by LMP
* Presenting symptoms: Bleeding score, Pain score
* USS Measurements: CRL, GS, RPOC 3 dimensions, Vascularity
* Discrepancy between gestation by CRL and LMP

All data will be collected retrospectively and annonymised.

Following data collection, machine learning models and feature reduction methods will be applied to determine the best performing model to predict success or failure of expectant or medical management of miscarriage respectively.

The next phase will include a prospective audit to collect data and test the predictive power of the MLM clinical decision support tool.

ELIGIBILITY:
Inclusion Criteria:

* Missed miscarriage and incomplete miscarriage less than 14weeks gestation
* Follow-up recorded at 2 weeks

Exclusion Criteria:

- Final outcome data unavailable

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases of missed miscarriage and incomplete miscarriage in the first trimester.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Machine learning predictive model development for miscarriage management outcomes. | Jan 2023- June 2024
  Machine learning predictive model development based on a retrospective audit of approximately 1000 cases of miscarriage.

SECONDARY OUTCOMES:
Prospective audit to test and validate predictive model | July 2024-June 2025
  To increase the sensitivity and specificity of the decision aid by widening the data collection to multiple sites and testing the machine learning model with prospective data.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Heatlhcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No